CLINICAL TRIAL: NCT07348484
Title: Diagnostic and Monitoring System for Chronic Kidney Disease Based on Urinary Biomarkers and Preventive Treatment With the SGLT2 Inhibitor Empagliflozin
Brief Title: Urinary Biomarker-Based Diagnostic and Monitoring System for Chronic Kidney Disease and Real-World Effectiveness of SGLT2 Inhibitors
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Other Study IDs: PI25/00053
Record Dates: First submitted 2025-11-18; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease
Keywords: SGLT2 inhibitors; empagliflozin; urinary biomarker
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Urine and plasma samples from patients included in the study, all of which will have chronic kidney disease and will be under treatment with empagliflozin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Empagliflozin Treatment Group: Participants with chronic kidney disease (CKD) stages 2-4 will receive oral empagliflozin (10-25 mg daily) for 12 months. Urinary and plasma samples will be collected at baseline, 6 months, and 12 months to evaluate the urinary biomarker panel, renal function (eGFR), and treatment safety.
  Interventions: Drug: Empagliflozin
- Control group: Adults with chronic kidney disease (CKD) stages 2-4 (KDIGO classification) managed in nephrology outpatient clinics without initiation of SGLT2 inhibitors at baseline or during follow-up.
  These patients receive standard clinical care according to local and national guidelines.
  They are followed on the same schedule (baseline, 6, and 12 months) and have identical variables collected from electronic health records and laboratory systems.
  Reasons for non-initiation of SGLT2i are documented systematically and may include:
  Not meeting indication criteria established by the Spanish National Health System (e.g., albumin-to-creatinine ratio <200 mg/g, eGFR <20 mL/min/1.73 m² for empagliflozin or <25 for dapagliflozin), or
  Clinical contraindications or conditions such as significant hypovolemia or hypotension, recurrent urinary or genital infections, or hypersensitivity.
  Control patients will be censored in the primary analysis if they later start SGLT2i therapy (cross-over).

INTERVENTIONS:
Drug: Empagliflozin — Oral empagliflozin (10-25 mg daily) for 12 months
  Groups: Empagliflozin Treatment Group

SUMMARY:
This prospective observational study aims to assess the association between real-world use of sodium-glucose co-transporter 2 inhibitors (SGLT2i; e.g., empagliflozin, dapagliflozin) and renal function decline in adults with chronic kidney disease (CKD) stages 2-4 (KDIGO classification). The study will also validate a urinary biomarker panel for early diagnosis and monitoring of CKD progression.

No investigational product is assigned, and medical practice or prescription patterns are not altered.

DETAILED DESCRIPTION:
This is a real-world, observational study with prospective follow-up and retrospective baseline data when available, conducted at the Nephrology Department of the University Hospital of Salamanca, Spain.

The project integrates translational and clinical components:

1. validation of a urinary biomarker panel obtained through differential proteomics for early detection and monitoring of CKD progression, and
2. evaluation of the effectiveness and safety of SGLT2i in routine clinical practice.

A total of 300 adults with CKD stages 2-4 will be included (150 initiating SGLT2i and 150 matched controls). Participants will be followed for 12 months (baseline, 6, and 12 months). Data will be extracted exclusively from electronic health records and laboratory systems.

The primary outcome is the annual decline rate of estimated glomerular filtration rate (eGFR, CKD-EPI 2021). Secondary outcomes include a composite renal endpoint (≥40% sustained eGFR decline, renal replacement therapy, transplantation, or renal death), cardiovascular hospitalization, all-cause mortality, adverse drug reactions (ADRs), and real-world patterns of SGLT2i use.

Exploratory analyses will assess associations between urinary biomarkers and clinical outcomes.

The study follows Spanish regulations for observational studies with medicinal products (Real Decreto 957/2020), with ethics approval and informed consent for biological samples.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Diagnosed with chronic kidney disease (KDIGO stages 2-4)
* Life expectancy ≥12 months
* Available clinical and laboratory data in the electronic medical record

Exclusion Criteria:

* Current or recent renal replacement therapy or kidney transplantation
* End-stage renal disease
* Participation in interventional trials that may affect outcomes
* Allergy or intolerance to SGLT2i (for exposed cohort)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with chronic kidney disease (CKD) stages 2-4.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in urinary biomarker panel expression (proteomic fingerprint) | Baseline, 6 months, 12 months
  Quantitative assessment of urinary biomarkers (including KIM-1, transferrin, IGFBP7, TIMP-2, among others) to evaluate disease progression and treatment response. Urinary biomarkers will be assessed using liquid chromatography-mass spectrometry (LC-MS/MS)-based differential proteomic analysis. Biomarker expression will be quantified as log2 fold change with false discovery rate (FDR) correction. Selected biomarkers will be validated using enzyme-linked immunosorbent assay (ELISA) or equivalent immunoassays. Biomarker concentrations will be normalized to urinary creatinine levels.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) | Baseline, 6 months, 12 months
  Evaluation of renal function improvement or stabilization during SGLT2 inhibitor treatment.
Histopathological improvement of renal tissue (animal study) | Monthly up to 9 months
  Monthly analysis of renal fibrosis, inflammation, and extracellular matrix accumulation in preclinical models treated with empagliflozin.
Monitoring of adverse events of empagliflozin in CKD patients without diabetes | From baseline to 12 months
  Adverse events (AEs) will be recorded and classified according to Common Terminology Criteria for Adverse Events (CTCAE, latest version), including severity grading and assessment of causality related to treatment.
  Serious adverse events (SAEs) and discontinuations due to AEs will be specifically tracked by the investigator.
Change in estimated glomerular filtration rate (eGFR) | From baseline to 12 months
  Change in renal function assessed by estimated glomerular filtration rate (eGFR) calculated using the CKD-EPI equation during empagliflozin treatment using the Serum creatinine-based CKD-EPI equation.
Change in serum creatinine | From baselinte to 12 months
  hange in serum creatinine levels to assess renal safety during treatment with empagliflozin by standard clinical laboratory assay (mg/dL).
Change in urinary albumin-to-creatinine ratio | From baseline to 12 months
  Change in urinary albumin-to-creatinine ratio as a marker of renal damage and safety during empagliflozin treatment by standard urine laboratory testing (mg/g creatinine).
Change in serum electrolyte levels | From baseline to 12 months
  Change in serum sodium and potassium levels to evaluate electrolyte safety during empagliflozin treatment by standard clinical laboratory testing (mmol/L).
Change in liver function tests | From baseline to 12 months
  Change in alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels to assess hepatic safety by standard clinical laboratory assays (U/L).
Change in glycated hemoglobin (HbA1c) | From baseline to 12 months.
  Change in HbA1c levels to monitor metabolic safety in non-diabetic CKD patients treated with empagliflozin by standard laboratory assay (%).
Change in hematological parameters | From baseline to 12 months
  Change in complete blood count parameters to evaluate hematological safety during treatment by standard clinical laboratory testing.
Change in blood pressure | From baseline to 12 months
  Assessment of changes in both blood pressures (systolic and diastolic), by Standard sphygmomanometer measurement (mmHg).
Change in body weight | From baseline to 12 months
  Change in body weight to assess tolerability and volume status during empagliflozin treatment by calibrated clinical scale (kg).
Discontinuation due to treatment intolerance | From baseline to 12 months
  Number and proportion of participants who permanently discontinue empagliflozin due to treatment-related intolerance or adverse events. It will be achieved trough clinical visit records and adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Martínez Salgado, PhD, Principal Investigator — University of Salamanca; Pilar Fraile Gómez, MD, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Hospital Universitario de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized datasets and analytic code will be available upon reasonable request, following approval by the Ethics Committee and IBSAL data governance board.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available starting 12 months after publication of primary results and for a minimum of 5 years thereafter.
Access Criteria: Qualified researchers with a methodologically sound proposal, as determined by the study steering committee, will be able to access the data. Requests should be directed to the study PI. A data access agreement will be required.